CLINICAL TRIAL: NCT01257763
Title: Tolerability Study of the Application of a 3M Microstructure Transdermal System by Finger Pressure to the Face in Healthy Subjects Stratified by Age and Fitzpatrick Skin Type
Brief Title: Tolerability Study of the Application of a 3M Microstructure Transdermal System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STU38370
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: needles/adverse effects; administration, cutaneous; erythema; pain measurement; Safety; Microstructure Transdermal System
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study device (Experimental): The study device is a transdermal microneedle array designed to introduce microscopic channels into the skin. The study device arm will receive application of this device.
  Interventions: Device: Transdermal Microchannel Skin System
- Sham device (Sham Comparator): The sham device will be very similar in appearance to the study device. The sham device arm will receive application of this device.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Transdermal Microchannel Skin System — A member of the research staff will apply the study device to the subject's lateral forehead, temple and nasolabial area on randomly selected sides of the face, 3 times at each anatomical location, for a total of 9 applications. All subjects will also receive 9 adjacent applications to the central forehead, and they will self-administer 3 adjacent applications to the chin under instruction of study staff.
  Arms: Study device
Device: Sham device — The side not receiving application of the study device at each anatomical location will receive a comparable number of applications of a sham device.
  Arms: Sham device

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of an experimental device that introduces microscopic channels into the skin. Creating microscopic channels in the skin allows for better absorption of various medications applied to the skin, and this study will determine if the study device offers a tolerable method by which to introduce these holes. The study population will include 54 individuals, ages 18-74 years old, with a roughly equal distribution of skin colors. Each subject will have a total of three visits 24 hours apart from one another. The study device will be applied at the Baseline and Day 1 visits. At various timepoints before and after device application, skin assessments for irritation will be completed using a 7-point Skin Reaction Scale and photographs will be taken. Subjects will report pain associated with device application using a standardized pain scale. At the baseline visit, a member of the research staff will administer applications of the study device on the side of the subject's forehead, temple and the area below and to the side of the nose on randomly selected sides of the face. The side of the face at each location not receiving application of the study device will receive applications of a "dummy" device. Subjects will not be informed of which device is the study device and which is the "dummy" device. At the Day 1 visit, a member of the research staff will administer study device applications to the center of the subject's forehead. The subject will also self-apply the study device to the chin, under the instruction of the research staff member. At the Day 2 visit, final skin assessments will be made and the subject will be evaluated and treated for any persistent skin irritation. Differences in skin irritation between sites of study device application and "dummy" device application will be determined, as well as several other endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-74 years old
* Subject in good health as determined by the investigator
* Subject has the willingness and the ability to understand and provide informed consent and communicate with the investigator

Exclusion Criteria:

* Subjects with active systemic or skin disease (including acne) or skin infection that could, in the opinion of the investigator, interfere with accurate study assessments
* Baseline skin irritation as defined by a local skin reaction score greater than "0" at any of the application areas (Appendix 1)
* Facial cosmetic procedures performed within 4 weeks of the baseline visit that may, in the opinion of the investigator, have an impact on skin assessment results†
* Topical medications applied to the face within 2 weeks of the baseline visit that may, in the opinion of the investigator, have an impact on skin assessment results†
* Subjects with skin disease such as atopic dermatitis, urticaria or dermatographism that may be exacerbated by device application †Subjects may enroll after a corresponding washout period

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Local skin reaction scores | 48 hours
  Difference in median local skin reaction scores between Study Device side and Control side for any of the three facial application sites at any of the seven follow-up times.
Median pain scores | 5 minutes
  Difference in median pain scores between Study Device side and Control side for any of the three facial application sites.
Local skin reaction and reported pain central forehead | 24 hours
  Reported pain and change in skin irritation at the central forehead site.
Local skin reaction score and reported pain chin | 24 hours
  Reported pain and change in skin irritation at the chin site.

SECONDARY OUTCOMES:
Max difference in skin reaction score | 48 hours
  Maximal difference in local skin reaction score at any follow-up visit
Subject questionnaire differences | 48 hours
  Reported differences in skin irritation or side-effects reported per patient questionnaire
Differences between skin type groupings | 48 hours
  Differences in reported pain or changes in local skin reaction score at central forehead site between the 3 Fitzpatrick skin type groupings (I-II, III-IV and V-VI).
Differences between age groups | 48 hours
  Differences in reported pain or changes in local skin reaction score at central forehead site between 3 age groupings (18-35, 36-60, 61-74).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P West, PhD, Study Director — Northwestern University; Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Hoesly FJ, Borovicka J, Gordon J, Nardone B, Holbrook JS, Pace N, Ibrahim O, Bolotin D, Warycha M, Kwasny M, West D, Alam M. Safety of a novel microneedle device applied to facial skin: a subject- and rater-blinded, sham-controlled, randomized trial. Arch Dermatol. 2012 Jun;148(6):711-7. doi: 10.1001/archdermatol.2012.280. PMID 22431712